CLINICAL TRIAL: NCT06303570
Title: A Single-Blind, Placebo-Control, Randomized Phase 2 Study to Evaluate the Efficacy and Safety of CBL-514 in Participants With Dercum's Disease Lipomas
Brief Title: A Study to Evaluate the Efficacy and Safety of CBL-514 Compared to Placebo in Participants With Dercum's Disease Lipomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBL-0202DD
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Dercum's Disease
Keywords: Adiposis Dolorosa; Lipedema; Lipomatosis; Skin Diseases; Lipid Metabolism Disorders; Metabolism Diseases; Connective Tissue Diseases
MeSH Terms: conditions — Adiposis Dolorosa; Lipedema; Lipomatosis; Skin Diseases; Lipid Metabolism Disorders; Connective Tissue Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBL-514 injection (Experimental): Eligible participants will receive CBL-514 administered in doses ranging from 1 mL to a maximum of 12 mL per lipoma, with treatments scheduled at intervals of approximately 4 weeks, up to 5 treatments.
  Interventions: Drug: CBL-514 injection
- 0.9% Sodium Chloride (Placebo Comparator): Eligible participants will receive 0.9% Sodium Chloride administered in doses ranging from 1 mL to a maximum of 12 mL per lipoma, with treatments scheduled at intervals of approximately 4 weeks, up to 5 treatments.
  Interventions: Drug: 0.9% Sodium chloride

INTERVENTIONS:
Drug: CBL-514 injection — The total injection volume per lipoma will based on the lipoma size,as determined by ultrasound. Dosing scheme is presented as below:
  Lipoma diameter of >0mm and <10mm - total injection volume per lipoma: 1 mL ; total of 5 mg CBL-514.
  Lipoma diameter of ≥10mm and ≤20mm - total injection volume per lipoma: 3 mL ; total of 15 mg CBL-514.
  Lipoma diameter of >20mm and ≤30mm - total injection volume per lipoma: 5 mL ; total of 25 mg CBL-514.
  Lipoma diameter of >30mm and ≤40mm - total injection volume per lipoma: 8 mL ; total of 40 mg CBL-514.
  Lipoma diameter of >40mm and ≤50mm - total injection volume per lipoma: 12 mL ; total of 60 mg CBL-514.
  Arms: CBL-514 injection
Drug: 0.9% Sodium chloride — The total injection volume per lipoma will based on the lipoma size,as determined by ultrasound. Dosing scheme is presented as below:
  Lipoma diameter of >0mm and <10mm - total injection volume per lipoma: 1 mL.
  Lipoma diameter of ≥10mm and ≤20mm - total injection volume per lipoma: 3 mL.
  Lipoma diameter of >20mm and ≤30mm - total injection volume per lipoma: 5 mL.
  Lipoma diameter of >30mm and ≤40mm - total injection volume per lipoma: 8 mL.
  Lipoma diameter of >40mm and ≤50mm - total injection volume per lipoma: 12 mL.
  Arms: 0.9% Sodium Chloride

SUMMARY:
This is a single-blind, placebo-controlled, randomized phase 2 study to evaluate the efficacy and safety of CBL-514 injections in participants with Dercum's Disease lipomas.

DETAILED DESCRIPTION:
This is a phase 2 study to evaluate the efficacy and safety of CBL-514 injections in participants with Dercum's disease lipomas.

A total of approximately 20 participants will be randomized. Eligible participants will be randomized (1:1) to receive either CBL-514 or placebo once every 4 weeks for up to 5 treatments for each selected lipoma. This means that there will be 10 participants in each dose group (CBL-514 group and placebo group). Eligible participants must have at least 4 and up to 10 painful individual lipomas. The injection volume per lipoma will depend on the lipoma size (as determined by ultrasound).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years to 64 years old (at screening), inclusive.
2. Body mass index (BMI) >18.5 kg/m2 at screening and Day 1.
3. Has confirmed DD and/or fulfills the following clinical criteria of DD in localized nodular form. The final diagnosis of disease is in the opinion of the Investigator.

   1. Chronic pain (>3 months) in the adipose tissue specific to the presence of lipomas and/or
   2. Pain in and around multiple lipomas.
4. Has at least 4 and up to 10 painful and well-defined lipomas with dimension of ≥10 mm and ≤50 mm as measured by ultrasound (read by the Investigator) at screening.
5. Generally considered healthy according to medical history, physical examination, ECG, and laboratory evaluation.
6. Voluntarily signs the informed consent form (ICF) and, in the opinion of the Investigator or designee, is physically and mentally capable of participating in the study, and willing to adhere to study procedures.

Exclusion Criteria:

1. Female participant of childbearing potential who is not willing to commit to an acceptable contraceptive regimen from the time of screening and throughout study participation until 90 days after the last IP dose, or who is currently pregnant or lactating. Female participant of childbearing potential who is breastfeeding or anticipates breastfeeding from the time of screening and throughout study participation until 90 days after the last IP dose. Male participant who is not willing to commit to using of a condom and refraining from sperm donation from the time of the first dose of IP, throughout study participation until 90 days after the last IP dose.
2. Unable to tolerate SC injections.
3. Diagnosed with another disorder with similar characteristics as DD as follows.

   1. Madelung's disease: multiple symmetric lipomatosis only localized in the upper body ie, shoulders, neck, or head.
   2. Panniculitis: inflammation of the SC adipose tissue, characterized by tender nodules and systemic signs.
   3. Proteus syndrome: disproportionate and asymmetric overgrowth of skin, and fatty and connective tissue.
   4. PTEN hamartoma syndrome: multiple hamartomas which includes segmental overgrowth, lipomatosis, arteriovenous malformation, and epidermal nevus.
   5. Gardner syndrome: multiple digestive adenomas with osteomas and multiple skin and soft tissue tumors.
4. Diagnosed with coagulation disorders or is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements, which inhibit coagulation or platelet aggregation.
5. Has fasting glucose concentration >200 mg/dL, delayed wound healing, bleeding risk, or any diabetic risks which, in the opinion of the Investigator or designee, is inappropriate to participate in the study.
6. Any clinically significant cardiac, hepatic, renal or neurologic/psychiatric disorders that in the opinion of the Investigator places the participant at significant risk, including but not limited to any of the following:

   1. Participants with cirrhosis or with inadequate liver function at screening defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, or total bilirubin >3.0 upper limit of normal (ULN).
   2. Participants with renal impairment, defined as both serum creatinine and blood urea nitrogen >1.5× ULN, or estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m2, or who are currently on dialysis.
7. Participant with a history of human immunodeficiency virus (HIV)-1 infection or participant with active HIV infection at screening with positive HIV antigen/antibody (Ag/Ab) combo test.
8. Participant is undergoing chronic steroid or immunosuppressive therapy, with the exception of:

   1. Use of oral steroid inhalation indicated for asthma management
   2. Use of topical steroid application for skin conditions that are not directly applied to or indirectly affect the treatment area
   3. Use of steroid as part of treatment for DD, and no side effects from chornic use.
9. Participant with active or prior history of malignancies within 5 years before screening or currently being evaluated for a possible malignancy, with the exception of adequately treated basal cell carcinoma of skin and in situ squamous cell carcinoma of skin at Investigator's discretion.
10. Abnormal skin, local skin conditions, or body modifications at the treatment area, which in the opinion of the Investigator, is inappropriate for participation in the study, including but not limited to any of the following:

    1. Prior wound, scar tissue, or infection in the treated area.
    2. Tattoo in the treated area.
11. Use of any analgesic except Cannabis within 2 days prior to Day 1 and use of Cannabis within 14 days prior to Day 1.
12. Requiring continual use of any medication that is known to strongly inhibit or induce CYP1A2 enzymes, sensitive CYP1A2 substrates or drugs with narrow therapeutic index during the study that, in the opinion of the Investigator, may affect the evaluation of the study product or place the participant at undue risk.
13. Participant who has undergone liposuction or aesthetic surgery to the region to be treated before screening or during the study, or aesthetic procedure for body contouring (eg, cryolipolysis, ultrasonic lipolysis, low level laser therapy, lipolysis injection) to the region to be treated within 12 months before screening or during the study.
14. Unable to receive local anesthesia.
15. Known allergies or sensitivities to the study drug or its components.
16. Use of other investigational drug or device within 12 weeks prior to screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To estimate the treatment effect, as measured by Partial Response (PR), between CBL-514 and placebo in participants with Dercum's disease (DD). | Week 20
  Lipoma volume will be determined by ultrasound assessment.

SECONDARY OUTCOMES:
To estimate the treatment effect, as measured by pain, between CBL-514 and placebo in participants with DD. | Week 20
  The Comparative Pain Scale is a 11-point scale (0-10) to assess pain from 0 being "pain free" to 10 being unimaginable/unspeakable pain.
To estimate the treatment effect, as measured by Complete Response (CR), between CBL-514 and placebo. | Up to 24 weeks
  Lipoma volume will be determined by ultrasound assessment.
To estimate the treatment effect, as measured by Partial Response (PR), between CBL-514 and placebo. | Week 24
  Lipoma volume will be determined by ultrasound assessment.
To evaluate the treatment effect, as measured by change in volume, between CBL-514 and placebo. | Up to 24 weeks
  Lipoma volume will be determined by ultrasound assessment.
To assess the treatment effect, as measured by pain, between CBL-514 and placebo. | Up to 24 weeks
  The Comparative Pain Scale is a 11-point scale (0-10) to assess pain from 0 being "pain free" to 10 being unimaginable/unspeakable pain.
To evaluate the incidence of adverse events of special interests (AESI) as defined in the protocol. | From baseline to 8 weeks post final treatment
  Adverse events (AEs) will be assessed by recording of clinical responses (e.g. treatment-emergent adverse events (TEAEs), and injection site reactions (ISRs)).
To evaluate the incidence of clinically significant abnormal findings as defined in the protocol as defined in the protocol. | From baseline to 8 weeks post final treatment
  Assessed by significant clinical changes in safety parameter (e.g. laboratory assessments, vital signs, ECGs, physical examinations).

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator Site, Spokane, Washington, United States